CLINICAL TRIAL: NCT03452371
Title: Hospital-based Patient Navigation to Promote Smoking Cessation: a Pilot Randomized Controlled Trial
Brief Title: Hospital-based Patient Navigation and Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-37040; 1UL1TR001430 (NIH)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Smoking Cessation
Keywords: Patient Navigation; Hospitalized smokers
MeSH Terms: conditions — Smoking Cessation | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Traditional Care (Active Comparator): Participants in this arm will receive usual care to help with smoking cessation offered to all patients who are smokers and some additional resources they can access for support.
  Interventions: Behavioral: Enhanced Traditional Care
- Patient Navigation Intervention (Experimental): Participants in this arm will meet with the trained patient navigator either in-person if she is available, or by telephone. They will receive up to ten hours of patient navigation over three months.
  Interventions: Behavioral: Patient Navigation

INTERVENTIONS:
Behavioral: Patient Navigation — Navigators will also screen participants for barriers to smoking cessation. Patient navigation intervention calls will use motivational interviewing (MI) strategies to: (1) Assess stage of change; (2) Assess and reinforce any prior abstinence from smoking and/or any efforts made to reduce/quit smoking; (3) Explore motivation to quit smoking, drawing on recent illness, financial/family situations as appropriate; advise about the risks of smoking and benefits of quitting (4) Discuss past experience with utilizing cessation support; (5) Explore potential barriers to using smoking cessation medications; (6) Brainstorm strategies to address identified barriers; (7) Elicit commitment to accept another patient navigation counseling call, discuss timing.
  Arms: Patient Navigation Intervention
Behavioral: Enhanced Traditional Care — Enhanced traditional care will include a resource card with information on quitlines, Boston Medical Center's (BMC's) Tobacco Treatment Center Program number, and websites for smoking cessation.
  Arms: Enhanced Traditional Care

SUMMARY:
In a pilot randomized controlled trial (RCT), smokers hospitalized on the general internal medicine or family medicine service will be randomized to: 1) enhanced traditional care (ETC), or 2) patient navigation (PN). Patients will be assessed at 3 months for self-report of quitting, use of smoking cessation medications, and use of counseling in the outpatient setting. Medical charts will be reviewed to ascertain if a prescription for smoking cessation medications was sent to the participants' pharmacy (primary outcome), if participants received inpatient tobacco counseling from the Tobacco Treatment Service (TTS), and whether they had a diagnosis of mental health and substance use.

DETAILED DESCRIPTION:
An Electronic Privacy Information Center(EPIC programmer who works with the Inpatient Tobacco Treatment Program will identify potential participants using electronic health record (EHR) data each week.

Eligible patients who are interested in the study and provide informed consent will be randomized and informed of the randomization assignment by the research assistant. We will stratify randomization by participants' response regarding their plan to quit smoking ("in the next month" or "more than a month from now"). A computer-generated sequence of random numbers will assign treatment groups. Participants will be randomized to one of two treatment arms: (1) standard of care, or (2) PN: a patient navigator to coordinate tobacco treatment with the smoker's outpatient healthcare team and address any underlying social determinants of health that are barriers to cessation (identified using a validated social determinants of health screening tool).

Assessments. A trained research assistant will administer these assessments either in-person or over the phone. The assessments require under 30 minutes to complete. The PI will also conduct an in-depth interview with the patient navigator to explore barriers to successful navigation. Outcome assessments will be conducted at baseline (prior to randomization) and at 3-months after randomization. Participants will be assessed at 3-months, for self-report of quitting, use of smoking cessation medications, and use of counseling in the outpatient setting.

Enhanced Traditional Care: Participants randomized to this group will receive a resource card that has information on quitlines, Boston Medical Center (BMC) outpatient program number, and websites for smoking cessation.

Patient Navigation Intervention: This intervention is based on the Social Contextual Model, a multi-level approach to health education which stresses the influence of life experiences (e.g. stress and financial problems) and social relationships (e.g. social networks and family roles) on the practice of health behaviors. Participants randomized into this group will meet the trained navigator in person if she is available, or will be introduced by telephone. Participants will receive up to ten hours of patient navigation, in person or over the phone, over a three-month period. Patient navigation contacts will involve individual counseling to help the patient achieve abstinence from smoking. Navigators will also screen participants for social determinants of health which may be preventing them from quitting smoking, using an adapted version of a validated social determinants of health screening tool. Patient navigation intervention calls will use motivational interviewing (MI) strategies to do the following: (1) Assess stage of change for smoking cessation; (2) Assess and reinforce any prior abstinence from smoking and/or any efforts made to reduce or quit smoking; (3) Explore the patient's motivation to quit smoking, drawing on recent illness, financial situation, and family situation as appropriate; advise about the risks of smoking and benefits of quitting (4) Discuss past experience with utilizing cessation support; (5) Explore potential barriers to using smoking cessation medications (e.g. lack of trust, cost, misconceptions about treatment (e.g. that nicotine replacement therapy (NRT) is more harmful than cigarettes); (6) Brainstorm strategies to address identified barriers; (7) Elicit commitment to accept another patient navigation counseling call, discuss timing.

Minimum navigation intervention dose: completion of social determinants of health screener and at least part of MI script (at least 1 item)

Navigator Training and Evaluation. A standard, validated motivational interviewing (MI) booster training program will be provided to one navigator. Training will include information about 1) tobacco dependence and treatment; and 2) barriers to treatment engagement among poor/minority patients. Our navigator will also be trained in MI. This additional training will take place over a half day and will focus on reviewing MI skills and delivery of the navigator intervention. MI skills will be reviewed through didactics, demonstrations, role-plays, and video. The navigator will be evaluated on both process (helpfulness, warmth, empathy), and content (intervention adherence). Following training the principal investigator (PI) will meet weekly with the navigator to ensure skill maintenance by reviewing audiotapes of intervention calls and providing corrective feedback.

Preserving Internal Validity/Treatment Fidelity, and Program Tracking. The intervention is manual-based. After each patient interaction, the navigator will complete a checklist of intervention components that were delivered. We will use these checklists to ensure that the intervention is delivered as intended, and to estimate intervention "dose" and treatment exposure. 5 participant interactions will be audio taped with permission from the participant. the PI will monitor tapes for protocol adherence.

Chart review. The research assistant will review participants' medical record to see if they have talked to their doctor about quitting smoking, if they have been prescribed medications to quit smoking, if they have attended a smoking cessation group at Boston Medical Center, if they received tobacco counseling from TTS, and if they have reduced the number of cigarettes or have quit smoking. We will collect data on mental health and substance use diagnoses. The investigators define mental health and substance use as the presence of diagnosed mental illness/substance use on the problem list/ annotations to problem list. the investigators will also determine whether participants have participated in any smoking cessation counseling sessions over the phone from the Massachusetts Quitworks Program.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Hospitalized on the General Internal Medicine or Family Medicine service
3. Have a primary care provider at BMC
4. Smoked ≥1 cigarettes/day in the past month
5. Must have plans to quit smoking
6. Read, understand, speak English
7. Possession of a telephone (home or cell)
8. Able to consent

Exclusion Criteria:

1. Cannot give informed consent or participate in counseling due to psychiatric or cognitive impairment or communication barrier
2. Admitted to surgical, obstetric or psychiatric units
3. Estimated life expectancy of <12 months
4. Medical instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Lasser, MD MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lasser KE, Quintiliani LM, Truong V, Xuan Z, Murillo J, Jean C, Pbert L. Effect of Patient Navigation and Financial Incentives on Smoking Cessation Among Primary Care Patients at an Urban Safety-Net Hospital: A Randomized Clinical Trial. JAMA Intern Med. 2017 Dec 1;177(12):1798-1807. doi: 10.1001/jamainternmed.2017.4372. PMID 29084312
- [Background] Lasser KE, Kenst KS, Quintiliani LM, Wiener RS, Murillo J, Pbert L, Xuan Z, Bowen DJ. Patient navigation to promote smoking cessation among low-income primary care patients: a pilot randomized controlled trial. J Ethn Subst Abuse. 2013;12(4):374-90. doi: 10.1080/15332640.2013.819311. PMID 24215228
- [Background] Kendzor DE, Businelle MS, Poonawalla IB, Cuate EL, Kesh A, Rios DM, Ma P, Balis DS. Financial incentives for abstinence among socioeconomically disadvantaged individuals in smoking cessation treatment. Am J Public Health. 2015 Jun;105(6):1198-205. doi: 10.2105/AJPH.2014.302102. Epub 2014 Nov 13. PMID 25393172
- [Background] Sorensen G, Barbeau E, Hunt MK, Emmons K. Reducing social disparities in tobacco use: a social-contextual model for reducing tobacco use among blue-collar workers. Am J Public Health. 2004 Feb;94(2):230-9. doi: 10.2105/ajph.94.2.230. PMID 14759932
- [Background] Borrelli B, McQuaid EL, Novak SP, Hammond SK, Becker B. Motivating Latino caregivers of children with asthma to quit smoking: a randomized trial. J Consult Clin Psychol. 2010 Feb;78(1):34-43. doi: 10.1037/a0016932. PMID 20099948
- [Background] Garg A, Butz AM, Dworkin PH, Lewis RA, Thompson RE, Serwint JR. Improving the management of family psychosocial problems at low-income children's well-child care visits: the WE CARE Project. Pediatrics. 2007 Sep;120(3):547-58. doi: 10.1542/peds.2007-0398. PMID 17766528
- [Background] Prochaska J, Redding C, Evers K. The Transtheoretical Model and Stages of Change. Health Behavior and Health Education: Theory, Research, and Practice.. Glanz K, Lewis FM, Rimer BK, editors. San Francisco: Jossey-Bass; 1997
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Traditional Care: Participants in this arm will receive usual care to help with smoking cessation offered to all patients who are smokers and some additional resources they can access for support.
  Enhanced Traditional Care: Enhanced traditional care will include a resource card with information on quitlines, BMC's Tobacco Treatment Center Program number, and websites for smoking cessation.
Period: Overall Study
Arm/Group | Enhanced Traditional Care | Patient Navigation Intervention
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Traditional Care | Patient Navigation Intervention | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (15) | 57 (10.1) | 54.9 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 13 | 6 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 3 | 6 | 9
  Non-Hispanic Black | 12 | 15 | 27
  Hispanic (any race) | 1 | 1 | 2
  Other/unknown | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 21 | 23 | 44
Intent to stop smoking [Count of Participants; unit: Participants]
  Within 30 days | 13 | 14 | 27
  Beyond 30 days | 8 | 9 | 17
Mean cigarettes per day [Mean (Standard Deviation); unit: cigarettes] | 11.3 (10.1) | 11.4 (10.4) | 11.4 (10.1)
Mean years smoked [Mean (Standard Deviation); unit: years] | 34.8 (18.2) | 39.9 (12.7) | 37.5 (15.5)
Mean Fagerstrom test score for nicotine dependence [Mean (Standard Deviation); unit: scores on a scale] — Standard validated 6 item instrument for assessing the intensity of addiction to nicotine. The 3 yes/no items are scored from 0 to 1. The 3 multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
  scores on a scale | 3.8 (2.8) | 3.7 (2.5) | 3.8 (2.6)
Mean quit attempt in past year [Mean (Standard Deviation); unit: quit attempts] | 1.7 (2.7) | 1.5 (1.7) | 1.6 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prescription for an FDA-approved Smoking Cessation Medication
Description: Based on chart review, whether a prescription for an FDA-approved smoking cessation medication was sent to the participants' pharmacy (Y/N)
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Traditional Care | Patient Navigation Intervention
Number analyzed (Participants) | 21 | 23
Participants | 9 | 11

2. Secondary Outcome: Number of Participants With Self-reported Smoking Cessation
Description: Self-report of 7-day point prevalence abstinence
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Traditional Care | Patient Navigation Intervention
Number analyzed (Participants) | 21 | 23
Participants | 1 | 2

3. Secondary Outcome: Number of Participants With Utilization of Smoking Cessation Medication
Description: self-report use of any smoking cessation medications (e.g. nicotine replacement therapy (NRT) patch, gum, lozenges, varenicline)
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Traditional Care | Patient Navigation Intervention
Number analyzed (Participants) | 21 | 23
Participants | 8 | 7

4. Secondary Outcome: Number of Participants With Stage of Change for Smoking Cessation
Description: Based on the Transtheoretical Model by Prochaska & DiClemente. The stages of change are: precontemplation, contemplation, preparation, action, maintenance, and relapse.
  Defined as moving from pre-contemplation to contemplation, or contemplation to preparation stage.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Traditional Care | Patient Navigation Intervention
Number analyzed (Participants) | 21 | 23
Participants | 3 | 4

5. Secondary Outcome: Mean Fagerstrom Test Score for Nicotine Dependence
Description: Standard validated 6 item instrument for assessing the intensity of addiction to nicotine. The 3 yes/no items are scored from 0 to 1. The 3 multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Enhanced Traditional Care | Patient Navigation Intervention
Number analyzed (Participants) | 12 | 14
scores on a scale | 1.9 (1.9) | 3 (2.6)

6. Secondary Outcome: Use of Other Tobacco Treatment Support
Description: Self-report of all tobacco treatment support received, including support from non-study sources, including the internet, during the 3-month study period.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Traditional Care | Patient Navigation Intervention
Number analyzed (Participants) | 21 | 23
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Enhanced Traditional Care | Patient Navigation Intervention
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 0/21 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03452371/Prot_SAP_000.pdf